CLINICAL TRIAL: NCT02687490
Title: A Prospective, Single-center, Open-Label, Phase II Study of Abraxane in Patients With Visceral Metastases Dominant Metastatic Breast Cancer
Brief Title: Abraxane in Patients With Visceral Metastases Dominant Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2016-20
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abraxane (Experimental): Abraxane: 125 mg/m2, D1, D8, D15 every 28 days
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — 125 mg/m2, D1, D8, D15

SUMMARY:
Abraxane in patients with visceral metastases dominant metastatic breast cancer

DETAILED DESCRIPTION:
A Prospective, Single-center, Open-Label, Phase II Study of Abraxane in patients with visceral metastases dominant metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic breast cancer;
2. Radiologically or histologically confirmed visceral dominant metastases;
3. Patients who are expected to acquire benefit from chemotherapy: ER and/or PR positive patients who developed resistance after prior endocrine therapy; HER2+ patients who experienced disease progression on prior target therapy and are not suitable for subsequent target therapy; mTNBC patients who relapsed after platinum therapy;
4. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1);
5. Patients who received paclitaxol in metastatic setting should be proven effective to prior paclitaxol based regimen and disease progressed after at least 3 months from the last administration of paclitaxol; those who received paclitaxel as neoadjuvant/adjuvant therapy can be enrolled if disease relapsed after at least 6 months from the completion of neoadjuvant/adjuvant chemotherapy. Patients who received docetaxol have no limitation for enrollment;
6. Eastern Cooperative Oncology Group performance (ECOG) status of 0-1;
7. All patients enrolled are required to have adequate hematologic, hepatic, and renal function;
8. Life expectancy longer than 12 weeks;
9. No medical history of serious cardiovascular, hepatic, respiratory or renal diseases;
10. Informed consent;
11. Patients with good compliance.

Exclusion Criteria:

1. Pregnant, lactating women or women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study;
2. Patients who are expected to acquire benefit from endocrine or target therapy;
3. Radiotherapy of axial bones within 4 weeks before enrollment or lack of recovery from prior radiotherapy;
4. Treatment with other experimental drug within 4 weeks before enrollment;
5. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to enrollment;
6. Other active malignancies (including other hematologic malignancies) or other malignancies within the last 5 years, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia;
7. Patients with a history of symptomatic cardiovascular, hepatic, respiratory, renal , hematological, endocrinal, neurological or psychiatric diseases;
8. Uncontrolled serious infection.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 8 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 8 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Xie Y, Gong C, Zhang J, Wang L, Cao J, Tao Z, Li T, Zhao Y, Li Y, Hu S, Wang B, Hu X. Phase II trail of nab-paclitaxel in metastatic breast cancer patients with visceral metastases. BMC Cancer. 2021 Nov 2;21(1):1174. doi: 10.1186/s12885-021-08921-2. PMID 34727875